CLINICAL TRIAL: NCT05162521
Title: The Impact of Lower Limb Fractures on Body Mass Index (BMI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kuwait Institute for Medical Specialization (Other Government)
Responsible Party: Principal Investigator, Ali Lari, Dr Ali Lari - MB BCh BAO, Kuwait Institute for Medical Specialization
Other Study IDs: KuwaitIMS2
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will prospectively follow patients with lower limb fractures to assess changes in weight after injury

ELIGIBILITY:
Inclusion Criteria:

* Adults with lower limb fractures

Exclusion Criteria:

* Polytrauma
* Upper limb fractures
* No consent
* Lack of follow up
* Patients opting for weight management treatments
* Patients with pre-existing mobility status impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with lower limb fractures
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
The impact of lower limb fractures on body mass index (BMI) | Change in weight over one year at different time intervals
  Assessing BMI at different time intervals after lower limb fractures

CONTACTS AND LOCATIONS:
Locations (1):
- AlRazi Orthopedic Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided